CLINICAL TRIAL: NCT01070810
Title: Thiamine as a Metabolic Resuscitator in Septic Shock
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Michael Donnino, Michael W. Donnino, MD, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2008P000053
Record Dates: First submitted 2010-02-17; First posted 2010-02-18 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-04

CONDITIONS: Septic Shock
Keywords: Septic Shock; Sepsis
MeSH Terms: conditions — Shock, Septic; Sepsis | interventions — Thiamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- 1 (Placebo Comparator): 50 ml D5W
  Interventions: Drug: D5W
- 2 (Experimental): 200mg Thiamine in 50ml D5W
  Interventions: Drug: Thiamine

INTERVENTIONS:
Drug: D5W — Dextrose 5%
  Arms: 1
Drug: Thiamine — Thiamine 200mg in 50ml D5W
  Arms: 2

SUMMARY:
The major goal of this project is to determine whether the use of thiamine in patients with septic shock will result in attenuation of lactic acidosis and a more rapid reversal of shock.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 18 years old
* Suspected or confirmed source of infection
* Hypotension (systolic pressure <90 mmHg) after a minimum 2 liter fluid bolus followed by vasopressor-dependence.
* Lactic Acidosis > 3 mmol/dl

Exclusion Criteria:

* Competing cause of lactic acidosis including: seizures within 3 hours of enrollment, use of linazolid metformin or anti-retrovirals at the time of enrollment, carbon monoxide or cyanide poisoning, highly suspected or known ischemic bowel, and known mitochondrial disorders
* Liver dysfunction specifically defined as AST or ALT elevation greater than 240
* Current Thiamine supplements or usage
* Competing indication for thiamine administration
* Cardiac Arrest
* DNR/DNI or comfort care status (DNR status in an intubated patient receiving full care is eligible)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2010-02; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael W Donnino, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Vine J, Lee JH, Kravitz MS, Grossestreuer AV, Balaji L, Leland SB, Berlin N, Moskowitz A, Donnino MW. Thiamine administration in septic shock: a post hoc analysis of two randomized trials. Crit Care. 2024 Feb 6;28(1):41. doi: 10.1186/s13054-024-04818-1. PMID 38321529

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: 50 ml D5W
  D5W: Dextrose 5%
- Thiamine: 200mg Thiamine in 50ml D5W
  Thiamine: Thiamine 200mg in 50ml Dextrose 5%
Period: Overall Study
Arm/Group | Placebo | Thiamine
Started | 45 | 43
Completed | 45 | 43
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Thiamine | Total
Number analyzed (Participants) | 45 | 43 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (17) | 70 (14) | 67 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 17 | 36
  Male | 26 | 26 | 52
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 40 | 36 | 76
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 45 | 43 | 88
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29 (7) | 29 (9) | 29 (8)

OUTCOME MEASURES:

1. Primary Outcome: Lactate Level 24 Hours After the First Study Medication Dose
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: mmol/L
Arm/Group | Placebo | Thiamine
Number analyzed (Participants) | 45 | 43
mmol/L | 2.6 [1.6 to 5.1] | 2.5 [1.5 to 3.4]
Statistical Analysis 1: Comparison: Placebo vs Thiamine; Test type: Superiority; p = 0.40, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Number of Participants With Shock Reversal
Description: Shock reversal was defined as > 24 hours off all vasopressors
Time Frame: Hospital stay, average 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Thiamine
Number analyzed (Participants) | 45 | 43
Participants | 32 | 32
Statistical Analysis 1: Comparison: Placebo vs Thiamine; Time to shock reversal was complicated by a high incidence of death prior to the event. To account for this we classified death as a competing risk event and used the estimated cumulative incidence function (CIF) to illustrate the comparison of CIFs between the two treatment groups using the Fine-Gray competing risk model. We tested the subdistribution hazards of these two CIF functions and obtained the estimated hazard ratio with 95% confidence intervals; Test type: Superiority; p = 0.97, Regression, Cox; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.61 to 1.62]

3. Secondary Outcome: APACHE II Score at 24 Hours
Description: APACHE II ("Acute Physiology and Chronic Health Evaluation II") is a severity-of-disease classification system; an integer score from 0 to 71 is computed based on several measurements; higher scores correspond to more severe disease and a higher risk of death
Time Frame: 24 hours
Population: APACHE II was not available on 6 patients in each group at 24 hour mostly because of early death.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Thiamine
Number analyzed (Participants) | 39 | 37
units on a scale | 26 (10) | 23 (8)
Statistical Analysis 1: Comparison: Placebo vs Thiamine; Test type: Superiority; p = 0.15, t-test, 2 sided

4. Other Pre Specified Outcome: Lactate Level at 24 Hours in Patients With Baseline Thiamine Deficiency
Description: Baseline thiamine deficiency was defined as a baseline thiamine level of ≤ 7 nmol/L
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: nmol/L
Groups:
- Thiamine Deficient Received Thiamine: Thiamine deficient (≤ 7 nmol/L) received 200mg Thiamine in 50ml D5W
- Thiamine Deficient, Received Placebo: Thiamine deficient (≤ 7 nmol/L) received 50ml D5W
Arm/Group | Thiamine Deficient Received Thiamine | Thiamine Deficient, Received Placebo
Number analyzed (Participants) | 15 | 13
nmol/L | 2.1 [1.4 to 2.5] | 3.1 [1.9 to 8.3]
Statistical Analysis 1: Comparison: Thiamine Deficient Received Thiamine vs Thiamine Deficient, Received Placebo; Test type: Superiority; p = 0.03, Wilcoxon (Mann-Whitney)

5. Other Pre Specified Outcome: Number of Participants Dying Before Hospital Discharge in Patients With Baseline Thiamine Deficiency
Description: Baseline thiamine deficiency was defined as a baseline thiamine level of ≤ 7 nmol/L
Time Frame: Hospital stay, average 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Thiamine Deficient Received Thiamine | Thiamine Deficient, Received Placebo
Number analyzed (Participants) | 15 | 13
Participants | 2 | 6
Statistical Analysis 1: Comparison: Thiamine Deficient Received Thiamine vs Thiamine Deficient, Received Placebo; Test type: Superiority; p = 0.10, Chi-squared

ADVERSE EVENTS:
Time Frame: Hospital stay, average 2 weeks
Arm/Group | Placebo | Thiamine
All-Cause Mortality (participants affected / at risk) | 19/45 | 19/43
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/43
Other Adverse Events (participants affected / at risk) | 0/45 | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No